CLINICAL TRIAL: NCT05702762
Title: Single Dose Aminoglycosides for Acute Uncomplicated Cystitis in the Emergency Department Setting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Health Ohio (Other)
Collaborators: Northeast Ohio Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-010
Record Dates: First submitted 2022-09-22; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Urinary Tract Infections
Keywords: gentamicin; single dose antibiotic treatment
MeSH Terms: conditions — Urinary Tract Infections | interventions — Gentamicins; Standard of Care; Cefdinir; Sulfamethoxazole; Trimethoprim; Time

STUDY DESIGN:
Intervention Model Description: Multicenter prospective open label randomized controlled study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gentamicin (Active Comparator): Subjects will be given one (1) injection intramuscular gentamicin 5 mg/kg (actual body weight unless patient is >120% ideal body weight in which case adjusted body weight will be utilized).
  Interventions: Drug: Gentamicin
- Standard of Care (Active Comparator): Oral antibiotic prescription
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Gentamicin — 5 mg/kg intramuscular injection
  Arms: Gentamicin
Drug: Standard of Care — Usual oral antibiotic multi-day dosing based on local antibiogram
  Other Names: Oral dose regimen for simple urinary tract infection: Including cephalexin, cefdinir, sulfamethoxazole/trimethoprim, and nitrofurantoin at appropriate dose, frequency, and duration
  Arms: Standard of Care

SUMMARY:
The purpose of this research study is to determine if gentamicin is as effective treatment of acute uncomplicated cystitis (urinary tract infection) using aminoglycosides versus the current standards of care. The current standards of care in our region are often to prescribe a multi-day antibiotic prescription that is taken multiple times per day whereas gentamicin will be a one-time dose in the emergency department. Gentamicin is the medicine being studied.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) account for more than 8 million office visits and 1 million emergency department visits each year in the United States, making them one of the most often encountered indications for antibiotic use in ambulatory care. Escherichia Coli has been shown to be the main cause of uncomplicated cystitis, occurring in 75-95% of cases, with other Enterobacteriaceae like Proteus mirabilis, Klebsiella pneumoniae and Staphylococcus saprophyticus comprising the majority of the other potential causes of cystitis. E. coli is also the most frequently encountered nitrite positive Enterobacteriaceae locally as well, representing nearly 3 out of every 4 culture specimens in the Boardman-specific gram-negative urine antibiogram (74%), 209 out of 284 to be exact. Some of the typical antibiotics used to treat these organisms had seen rising resistance rates from 2003-2012, with substantial increases in the resistance to both ciprofloxacin (3.6% to 11.8%) and trimethoprim-sulfamethoxazole (17.2% to 22.2%) in the United States. Gentamicin offers 93% sensitivity towards E. coli in the local antibiogram, whereas sulfamethoxazole-trimethoprim and fluoroquinolones offer 75% and 69%, respectively. More importantly, the current standard of care, cefdinir, only offers around 80% sensitivities locally. While nitrofurantoin has retained high levels of antibiotic activity against E. coli, it is contraindicated in the elderly and patients with poor renal function. This growing rate of resistance has placed a larger emphasis on finding alternative treatment options.

As stated above, Goodlet et al. reviewed 13 studies totaling 13,804 patients, and data from 11 out of the 13 revealed a microbiological cure rate of 94.5% +/- 4.3% using single dose aminoglycosides to treat urinary tract infections. Seven of these studies had comparator groups that included medications such as oral cephalosporins, Fosfomycin, trimethoprim-sulfamethoxazole and amoxicillin. No difference in initial or sustained microbiological cure rate in those that received aminoglycosides versus other medications was demonstrated. Only two of the thirteen studies evaluated clinical cure rates which were shown to be 82.8% and 94.7%, respectively. In the studies with 30 day follow up, an overall recurrence rate at 30 days was found to be 19% (84/443 patients). The recurrence rate seen using aminoglycosides is improved when compared to the general population, as 27% of women have been found to experience recurrence of their symptoms within 6 months of having urinary tract infections. Aminoglycosides were at one time a standard first-line therapeutic option to treat UTIs but fell out of favor due to their side effect profile.

The most concerning adverse effects of aminoglycosides were mainly seen in association with multi-day regimens of the drugs. Their nephrotoxic and ototoxic effect are seen in less than 1% of patients evaluated, but saw their use decrease roughly 41% between 2002-2009. In the Goodlet et al. study only 63 of the 13,804 patients (0.5%) reported adverse effects associated with the single dose aminoglycoside treatment. Only 7 total cases (0.05%) reported nephrotoxicity and 53 total cases (0.38%) reported signs of vestibular toxicity such as tinnitus and equilibrium disorders. Additionally, in a study of over 10,000 patients receiving single dose amikacin for UTI, nephrotoxicity was only reported in 0.04% of cases. Another review looking at 24,107 patients that had received a single dose of gentamicin reported no cases of ototoxicity as well. Comparably, sulfamethoxazole-trimethoprim carries common and rare risks of hyperkalemia, blood dyscrasias, hypersensitivity reactions, and other adverse events affecting nearly every organ system of the body. Fluoroquinolones carry common and rare risks of QT segment prolongation, peripheral neuropathy, dysglycemia, adverse events affecting the whole body and even a long-term syndrome effecting tens of thousands of people called fluoroquinolone-associated disability (FQAD). Beta-lactams such as cefdinir commonly cause gastrointestinal symptoms but more rarely effect other organ systems such as the skin, metabolic and hematologic abnormalities, and other adverse events as well. While adverse effects may occur with aminoglycosides, the studied risk of single dose use is not extreme and comparable with adverse effects seen with current standards of care.

While there is a proven cure rate utilizing single dose aminoglycosides to treat acute uncomplicated cystitis, they will also provide several other benefits when used in the emergency department setting. The single dosing of antibiotic in the emergency department removes the need for patient adherence to outpatient antibiotic therapy, thus reducing possible bounce back visits. Gentamicin can also be administered intramuscularly, as it was in all the above studies, both removing the need for IV access and expediting possible disposition in the emergency department. Lastly, greater than 75% of outpatient UTI prescriptions are written for durations that are not recommended, which is an issue that can be removed from the equation entirely utilizing single dose treatment. Treating patients with single dose aminoglycosides for acute uncomplicated cystitis in the emergency department may provide better compliance with the same efficacy, resulting in a new standard of care for treatment in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, woman, pre-menopausal, non-pregnant with clinical signs of urinary tract infection and nitrite positive urine.

Exclusion Criteria:

* Contraindications include hypersensitivity to gentamicin or other aminoglycosides.
* Patients younger than 18 years of age.
* Pregnant or post-menopausal patients.
* Patients without symptoms of UTI, nitrite negative urine, or any patient with working diagnosis of complicated UTI such as pyelonephritis or any patient catheterized.
* ANY history of pre-existing renal impairment.
* Patient that has any listed or reports taking ANY nephrotoxic or wit drug-drug interaction medication in the past 7 days (see Appendix 5).
* ANY history of hearing loss, tinnitus, or vertigo.
* ANY patient that has received general anesthesia or neuromuscular blockade in past 7 days.
* Patients with ANY history of neuromuscular disorders including: myasthenia gravis, amyotrophic lateral sclerosis, muscular dystrophy, botulism, congenital myasthenic syndromes, congenital myopathies, myositis, Lambert-Eaton syndrome, mitochondrial myopathy, myotonic dystrophy, neuromyotonia, or peripheral neuropathy.
* Patients with ANY history of thrombocytopenia.
* Patient that has any listed or reports taking ANY anticoagulants in the past 7 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Resolution | 7 days from presentation
  If patient is or is not still having any pain with urination, urinary frequency or urinary urgency
Clinical Resolution | 30 days from presentation
  If patient is or is not still having any pain with urination, urinary frequency or urinary urgency

CONTACTS AND LOCATIONS:
Locations (1):
- St. Elizabeth Youngstown Hospital, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodlet KJ, Benhalima FZ, Nailor MD. A Systematic Review of Single-Dose Aminoglycoside Therapy for Urinary Tract Infection: Is It Time To Resurrect an Old Strategy? Antimicrob Agents Chemother. 2018 Dec 21;63(1):e02165-18. doi: 10.1128/AAC.02165-18. Print 2019 Jan. PMID 30397061
- [Background] Durkin MJ, Keller M, Butler AM, Kwon JH, Dubberke ER, Miller AC, Polgreen PM, Olsen MA. An Assessment of Inappropriate Antibiotic Use and Guideline Adherence for Uncomplicated Urinary Tract Infections. Open Forum Infect Dis. 2018 Aug 10;5(9):ofy198. doi: 10.1093/ofid/ofy198. eCollection 2018 Sep. PMID 30191156
- [Background] Ababneh M, Harpe S, Oinonen M, Polk RE. Trends in aminoglycoside use and gentamicin-resistant gram-negative clinical isolates in US academic medical centers: implications for antimicrobial stewardship. Infect Control Hosp Epidemiol. 2012 Jun;33(6):594-601. doi: 10.1086/665724. Epub 2012 Apr 19. PMID 22561715
- [Background] Foxman B. The epidemiology of urinary tract infection. Nat Rev Urol. 2010 Dec;7(12):653-60. doi: 10.1038/nrurol.2010.190. PMID 21139641
- [Background] Kang CI, Kim J, Park DW, Kim BN, Ha US, Lee SJ, Yeo JK, Min SK, Lee H, Wie SH. Clinical Practice Guidelines for the Antibiotic Treatment of Community-Acquired Urinary Tract Infections. Infect Chemother. 2018 Mar;50(1):67-100. doi: 10.3947/ic.2018.50.1.67. PMID 29637759
- [Background] Sanchez GV, Babiker A, Master RN, Luu T, Mathur A, Bordon J. Antibiotic Resistance among Urinary Isolates from Female Outpatients in the United States in 2003 and 2012. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2680-3. doi: 10.1128/AAC.02897-15. Print 2016 May. PMID 26883714
- See also: . International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women — https://academic.oup.com/cid/article/52/5/e103/388285